CLINICAL TRIAL: NCT04728308
Title: Does Bupivacaine Infiltration Reduce Postoperative Pain in Patients With Cesarean Section?
Brief Title: Bupivacaine Infiltration and Postoperative Pain
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, Dr Arshad Khushdil, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A/28/EC/232/2021
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Local Infiltration; Analgesia
Keywords: Bupivacaine; Local anesthetic; cesarean section
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Informed written consent will be taken. Patients will be divided into two groups randomly, by a computer-generated method. Caesarean section will be done under spinal anesthesia by a well-trained consultant obstetrician. The surgeon will be provided with a 20 ml syringe filled either with 20 ml of 0.5% Bupivacaine or 20 ml of placebo (distill water). The syringe will be prepared by our researcher obstetrician. The contents of the syringe will be determined by numbers generated from the computer and the operating surgeon will be unaware of these contents. Before closing the skin incision, the operating surgeon will infiltrate the solution in subcutaneous tissue around the incision.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Caesarean section will be done under spinal anesthesia by a well-trained consultant obstetrician. The surgeon will be provided with a 20 ml syringe filled either with 20 ml of 0.5% Bupivacaine or 20 ml of placebo (distill water). The syringe will be prepared by our researcher obstetrician. The contents of the syringe will be determined by numbers generated from the computer and the operating surgeon will be unaware of these contents. Before closing the skin incision, the operating surgeon will infiltrate the solution in subcutaneous tissue around the incision. Severity of pain , need for amount of opioids and duration of hospital stay will be assesed by doctor incharge in postoperative ward.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): 20ml of 0.5% bupivacaine is infiltrated in the subcutaneous tissue around the incision site
  Interventions: Drug: Bupivacain
- Placebo group (Placebo Comparator): 20 ml of distill water is infiltrated in the subcutaneous tissue around the incision site
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — Before closing the skin incision,Infiltration of 20ml of 0.5% bupivacaine around incision site will be done in the patients of experimental group and 20 ml of distill water will be infiltrated in the pateints of the placebo group

SUMMARY:
This is a double-blind randomized controlled trial to assess the efficacy of local infiltration of bupivacaine versus placebo, in reducing postoperative pain. The severity of pain will be assessed in terms of mean score on visual analogue scale, opioid requirement and average duration of hospital stay.

DETAILED DESCRIPTION:
Objective: To compare the effect of bupivacaine wound infiltration with placebo during caesarean section in terms of mean pain scores, analgesic requirement, and duration of hospital stay

Introduction:

Over the last several decades, the rate of caesarean has increased rapidly.According to the data collected from 150 countries, almost 18.6% of the total births occur by caesareansection, with rates ranging from 6% to 27% in different regions. In Egypt and Turkey, the rate of caesarean section is more than 50%. In Pakistan, caesarean section rate was found to be 15.8% in 2013, with a rate of 11.5% in rural areas and 25.6% in the urban population.

Caesarean section is the most commonly performed surgical procedure nowadays and is associated with moderate to severe pain after the surgery. Pain after caesarean section occurs due to inadvertent damage to parietal peritoneum and nerve supply of skin.According to a survey done in America in 2003, it was found that upto 70% of the patients will experience severe pain postoperatively. Severe pain after caesarean section specifically affects mother-baby bonding, lactation, and patient recovery. It also leads to a prolonged hospital stay, reduced mobility, and consequently increasing the risk of thromboembolic disease in the postoperative period. Severe pain aftercaesarean delivery has also been found to be associated with postnatal depression and pain persisting after 8 weeks of delivery.Incaesarean delivery, the provision of effective postoperative analgesia is of key importance to facilitate early ambulation and infant care. It is also very important that the type of analgesia providedis safe, effective,and has minimal side effects for the mother and her baby.

The most appropriate method of analgesia for postoperative pain after caesarean section remains uncertain.Different methods have been used for this purpose. Parenteral opioids are the most commonly used method but associated nausea, vomiting, sedation, and risk of respiratory depression in mother and baby limits its use. Continuous epidural analgesia or patient-controlled analgesia also provide effective analgesia and have fewer adverse effects butare expensive and require special equipment and expertise.Infiltration of local anesthetic into subcutaneous tissue around the incision site has also been thought to relieve pain after caesarean section. Local anesthetic drugslike lignocaine and bupivacaine inhibit nerve impulses from the site of injury thus providing an analgesic effect. However,in this regard, there is no consistent evidence.Some studies show high efficacy while others report no benefit.

This study is being conducted to assess the effectiveness of wound infiltration of 20ml of 0.5% bupivacaine after the caesarean section on postoperative pain scores and analgesic requirement. If found effective this regimen can be implemented locally as it is cheap and simple to use.

Method: This will be a a double-blind randomized controlled trial. It is being conducted at the Department of Gynecology and Obstetrics, Pak Emirates Military Hospital from 10th January 2020 and will be completed till 10th april 2021. Pregnant women at term, with ages between 20 to 40 years, who are planned to undergo elective caesarean section, will included in the study. Patients are divided into two groups by a computer-generated lottery method. In group A, 20 ml of sterile water is infiltrated in the subcutaneous tissue around the incision site while 20 ml of 0.5% bupivacaine injection is infiltrated in patients of group B. The primary outcome measure is to asses the difference in postoperative pain among the two groups in terms of average pain score measure with help of visual analogue scale (VAS) and total dose of analgesia required in the first twenty four hours after the surgery. Secondary outcome is the average duration of hospital stay in patients of the two groups All the data will be entered and analyzed with help of SPSS version 16. For quantitative variables like mean pain score, average dose of opioid required, and average duration of hospital stay, the investigators will calculate mean and standard deviation and for qualitative variables like indication of the caesarean section, frequency and percentage will be calculated. To compare the quantitative variables between the two groups, unpaired T-test and for comparison of qualitative variables, chi-square test will be used. A p-value of <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with age between 20-40 years, American Society of Anesthesiologist (ASA) class II, BMI < 35 at the time of surgery, a period of gestation 37+0- 40+0 weeks, elective caesarean section done under spinal anesthesia, skin incision pfennensteil and lower segment transverse incision on the uterus.

Exclusion Criteria:

* allergy to local anesthetic, emergency caesarean section, conversion of spinal anesthesia to general anesthesia, caesarean section due to abnormal placentation, midline skin incision, upper segment incision on uterus

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-04-10 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
average pain score on Visual analogue scale | in first 12 hours after the surgery
  average pain score on Visual analogue scale in first 12 hours after the surgery
average opioid consumption | within first 24 hours after the surgery
  average consumption of tramadol injection

SECONDARY OUTCOMES:
average duration of hospital stay | 3 months
  average duration of hospital stay after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Madiha Ahmed, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No